CLINICAL TRIAL: NCT05625243
Title: Evaluation of the Proximal Contact Quality in Posterior Complex Carious Cavities Restored With Bulk Fill Ormocer and Resin Composite Using a Precontoured Circumferential Matrix System Versus Precontoured Sectional Matrix System
Brief Title: Evaluation of the Proximal Contact Quality in Posterior Complex Carious Cavities Restored With Bulk Fill Ormocer and Resin Composite Using a Precontoured Circumferential Matrix System Versus Pre Contoured Sectional Matrix System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Alghaffar Khafagi, Evaluation of the proximal contact quality in posterior complex carious cavities restored with bulk fill ormocer and resin composite using a precontoured circumferential matrix system versus precontoured sectional matrix system, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14422018454217
Record Dates: First submitted 2022-11-10; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Posterior Complex Carious Proximal Cavities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bulk-fill ormocer with Precontoured circumferential matrix system (Experimental): A suitable size precontoured circumferential matrix band will be selected and placed. Teeth separation will be acquired with a suitable size wedge and a separation ring . Then the bulk-fill ormocer will be applied and light cured according to the manufacturer instructions.
  Interventions: Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA); Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured sectional matrix systym (Saddle matrix, TORVM, Moscow, Russia); Other: Bulk-fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA)
- Bulk-fill ormocer with Precontoured Saddle matrix system (Experimental): Teeth separation will be acquired with a suitable size wedge (fixing wooden wedges and a separation ring Then the bulk-fill ormocer will be applied and light cured according to the manufacturer instructions.
  Interventions: Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA); Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured sectional matrix systym (Saddle matrix, TORVM, Moscow, Russia); Other: Bulk-fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA)
- X-tra fill, Voco) with Precontoured circumferential matrix (Palodent 360, Dentsply ) (Experimental): .Bulk-fill resin composite (X-tra fill, Voco) with Precontoured circumferential matrix system (Palodent 360) will be applied
  Interventions: Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA); Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured sectional matrix systym (Saddle matrix, TORVM, Moscow, Russia); Other: Bulk-fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA)
- Bulk-fill resin composite with Precontoured sectional matrix systym (Active Comparator): Teeth separation will be acquired with a wooden wedge and a separation ring (Delta ring, TORVM, Moscow, Russia). Then the bulk fill resin composite will be applied and light cured according to the manufacturer instructions.
  Interventions: Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA); Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured sectional matrix systym (Saddle matrix, TORVM, Moscow, Russia); Other: Bulk-fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA)

INTERVENTIONS:
Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA) — A suitable size precontoured circumferential matrix band (Palodent 360, Dentsply Caulk, Millford DE, USA) will be selected and placed. Teeth separation will be acquired with a suitable size wedge (Palodent V3, Dentsply Caulk, Millford DE, USA) and a separation ring (Palodent V3 universal ring, Dentsply Caulk, Millford DE, USA). Then the bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) will be applied and light cured according to the manufacturer instructions.
Other: Bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) with Precontoured sectional matrix systym (Saddle matrix, TORVM, Moscow, Russia) — A suitable size precontoured sectional matrix band (Saddle matrix, TORVM, Moscow, Russia) will be selected and placed. Teeth separation will be acquired with a suitable size wedge (fixing wooden wedges, TORVM, Moscow, Russia) and a separation ring (Delta ring, TORVM, Moscow, Russia). Then the bulk-fill ormocer (Admira fusion x-tra, Voco, Cuxhaven, Germany) will be applied and light cured according to the manufacturer instructions.
Other: Bulk-fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) with Precontoured circumferential matrix system (Palodent 360, Dentsply Caulk, Millford DE, USA) — A suitable size precontoured circumferential matrix band (Palodent 360, Dentsply Caulk, Millford DE, USA) will be selected and placed. Teeth separation will be acquired with a suitable size wedge (Palodent V3, Dentsply Caulk, Millford DE, USA) and a separation ring (Palodent V3 universal ring, Dentsply Caulk, Millford DE, USA). Then the bulk fill resin composite (X-tra fill, Voco, Cuxhaven, Germany) will be applied and light cured according to the manufacturer instructions.

SUMMARY:
The use of ormocers with precontoured circumferential matrix system allow predictable restoration of complex proximal posterior cavities with less time and fewer tools required to produce optimum proximal contact size, location and magnitude and restoration durability with higher wear resistance.

DETAILED DESCRIPTION:
After profound local anesthesia, conservative cavity preparations will be performed with high-speed burs (no.:330, Meisinger, Germany) under constant refrigeration. Intermittent rotary instrument contact with tooth limited to the removal of compromised enamel. The cavity outline is restricted to the removal of carious tissue with spherical carbide burs at low speed. In the removal of defective restorations, the friable enamel and remnant carious tissue will be removed in the same way. All teeth will be restored using a rubber dam. The universal bonding agent (Voco, Cuxhaven, Germany) will be applied with previous selective enamel etching with 37% phosphoric acid for 30 seconds. These materials will be inserted following the manufacturer's instructions.

After cavity preparation, each participant will choose a random number from an opaque sealed envelope, then patient will select from random numbers prepared by Y.H. to randomly assign interventions to the participant oral cavity.

All restorations will be prepared, restored, finished and polished by one operator.

ELIGIBILITY:
Inclusion Criteria:

- Posterior complex proximal carious lesions Vital upper or lower posterior teeth with no signs of irreversible pulpitis. Presence of adjacent and opposing teeth with normal occlusion

Exclusion Criteria:

* Proximal carious cavities in the mesial surface of first premolars. Periapical pathology or signs of pulpal pathology. Possible prosthodontic restoration of teeth. Heavy occlusion and occlusal contacts or history of bruxism. Pulpitis, non-vital or endodontically treated teeth. Sever periodontal affection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-11-26 (Estimated); Primary Completion 2023-11-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proximal Contact quality | one year follow up
  50 micro sectional matrix band (Saddle matrix, TORVM, Moscow, Russia)
  FDI criteria (Hickel et al., 2010)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alghaffar khafagi, master, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University,, Cairo, Egypt